CLINICAL TRIAL: NCT03234816
Title: Vasopressor Prophylaxis After Spinal Anesthesia: A Dose Finding Study
Brief Title: Vasopressor Prophylaxis After Spinal Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Principal investigator, Lecturer of anesthesia and critical care medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: N_66_2017
Record Dates: First submitted 2017-07-27; First posted 2017-07-31 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — Norepinephrine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- - 0.05 mcg /Kg/min group (Experimental): will receive norepinephrine 0.05 mcg /Kg/min after spinal anesthesia by bupivacaine till five-minutes after delivery of the fetus
  Interventions: Drug: Norepinephrine 0.05 mcg /Kg/min; Drug: Bupivacaine
- - 0.1 mcg /Kg/min group (Experimental): will receive norepinephrine 0.1 mcg /Kg/min after spinal anesthesia by bupivacaine till five-minutes after delivery of the fetus
  Interventions: Drug: Norepinephrine 0.1 mcg /Kg/min; Drug: Bupivacaine
- - 0.15 mcg /Kg/min group (Experimental): will receive norepinephrine 0.15 mcg /Kg/min after spinal anesthesia by bupivacaine till five-minutes after delivery of the fetus
  Interventions: Drug: Norepinephrine 0.15 mcg /Kg/min; Drug: Bupivacaine

INTERVENTIONS:
Drug: Norepinephrine 0.05 mcg /Kg/min — Norepinephrine infusion by rate of 0.05 mcg /Kg/min after spinal anesthesia
  Other Names: noradrenaline infusion
  Arms: - 0.05 mcg /Kg/min group
Drug: Norepinephrine 0.1 mcg /Kg/min — Norepinephrine infusion by rate of 0.05 mcg /Kg/min after spinal anesthesia
  Other Names: noradrenaline infusion
  Arms: - 0.1 mcg /Kg/min group
Drug: Norepinephrine 0.15 mcg /Kg/min — Norepinephrine infusion by rate of 0.05 mcg /Kg/min after spinal anesthesia
  Other Names: noradrenaline infusion
  Arms: - 0.15 mcg /Kg/min group
Drug: Bupivacaine — 10 mg Bupivacaine intra-thecal for spinal anesthesia
  Other Names: marcaine

SUMMARY:
Norepinephrine has been recently introduced as a prophylactic vasopressor during Cesarean delivery with promising results ; However, the optimum dose for efficient prophylaxis with the least side effects is not known. In this study, we will compare three doses (0.05, 0.1, 0.15 mcg/Kg/min) of norepinephrine for prophylaxis against Post-Spinal hypotension during cesarean delivery.

DETAILED DESCRIPTION:
Maternal hypotension is a common complication after spinal anesthesia for cesarean delivery (CD). Using vasopressors have been considered a gold standard for prevention of post-spinal hypotension (PSH) during CD.

Norepinephrine (NE) is a potent vasopressor characterized by both α adrenergic agonistic activity in addition to a weak β adrenergic agonistic activity; thus, NE is considered a vasopressor with minimal cardiac depressant effect; these pharmacological properties would make NE an attractive alternative to phenylephrine and ephedrine (the most commonly used vasopressors in obstetric anesthesia).

Norepinephrine has been recently introduced as a prophylactic vasopressor during CD with promising results; However, the optimum dose for efficient prophylaxis with the least side effects is not known.

In this study, we will compare three doses (0.05, 0.1, 0.15 mcg/Kg/min) of norepinephrine for prophylaxis against PSH during CD.

ELIGIBILITY:
Inclusion Criteria:

* full term singleton pregnant women
* Scheduled for elective Cesarean Delivery
* Aged between 18 and 40 years

Exclusion Criteria:

* Cardiac morbidities
* Hypertensive disorders of pregnancy,
* Peripartum bleeding
* Baseline systolic blood pressure (SBP) < 100 mmHg
* Body mass index > 35

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 270 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
incidence of postspinal hypotension | 30 minutes after spinal anesthesia
  The number of patients who develop hypotension (defined as decreased SBP less than 80% of the baseline reading during the period from intrathecal injection till delivery of the fetus) after spinal block divided by the total number in the group

SECONDARY OUTCOMES:
heart rate | 90 minutes after spinal anesthesia
  heart rate after spinal anesthesia measured in beat per minute
vomiting | 120 minutes after spinal anesthesia
  incidence of vomiting after spinal anesthesia
nausea | 120 minutes after spinal anesthesia
  incidence of nausea after spinal anesthesia
ephedrine consumption | 60 minutes after spinal anesthesia
  total amount of ephedrine consumed after spinal anesthesia
Atropine consumption | 60 minutes after spinal anesthesia
  total amount of atropine consumed after spinal anesthesia
APGAR score | 10 minutes after delivery
  APGAR score of the delivered fetus
incidence of severe postspinal hypotension | 30 minutes after spinal anesthesia
  The number of patients who develop hypotension (defined as decreased SBP less than 60% of the baseline reading during the period from intrathecal injection till delivery of the fetus) after spinal block divided by the total number in the group
arterial blood pressure | 90 minutes after spinal anesthesia
  arterial blood pressure after spinal anesthesia measured in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mukhtar, Professor, Study Director — Head of research committee section in anesthesia department
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No